CLINICAL TRIAL: NCT04958447
Title: Nutritional Management in Respiratory Critically Ill Patients -an Observational Study in Mainland China
Acronym: NM-in-RCIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Longyan First Affiliated Hospital of Fujian Medical University (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Peking University International Hospital (Other); Peking University People's Hospital (Other); Peking University Shougang Hospital (Other); Beijing Jingmei Group General Hospital (Unknown); Beijing Fangshan District Liangxiang Hospital (Other); Beijing Hospital (Other Government); Beijing Coal Group General Hospital (Unknown); Beijing Rehabilitation Hospital (Other); Beijing 302 Hospital (Other); Cangzhou People's Hospital (Other); Cangzhou Central Hospital (Other); Affiliated Hospital of Chengde Medical University (Other); Huan'an First People's Hospital (Other); The First Affiliated Hospital of Hebei North University (Other); Hebei Sheng Xiong Ke Yi Yuan (Unknown); The Second Hospital of Hebei Medical University (Other); North China University of Science and Technology (Other); First Hospital of Shijiazhuang City (Other); Tangshan Central Hospital (Other); Zhuozhou Hospital (Unknown); Second Hospital of Jilin University (Other); The First Hospital of Jilin University (Other); The General Hospital of Northern Theater Command (Other); Affiliated Zhongshan Hospital of Dalian University (Other); Dalian Municipal Central Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Central Hospital Affiliated to Shenyang Medical Collage (Other); The Fourth Affiliated Hospital of China Medical University (Other); First Hospital of China Medical University (Other); Tianjin Medical University General Hospital (Other); Tianjin Chest Hospital (Other); Tianjin Medical University Second Hospital (Other); Special Medical Center of the Armed Police Force (Unknown); The Second People Hospital of Wuhu (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Meizhou People's Hospital (Other); The General Hospital of Southern Theater Command (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Hainan People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The General Hospital of Eastern Theater Command (Other); Huai an First People Hospital (Unknown); Subei People's Hospital of Jiangsu Province (Other); The First People's Hospital of Lianyungang (Other); Nanjing No.1 Hospital (Unknown); The Affiliated Jiangning Hospital of Nanjing Medical University (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Soochow University (Other); Suzhou Municipal Hospital (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); Jiangxi Provincial People's Hopital (Other); Second Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Nanchang University (Other); Shaanxi Provincial People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xijing Hospital (Other); Sichuan Provincial People's Hospital (Other); No.2 People Hospital of Fuyang City (Unknown); The Second Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Tongji Hospital (Other); Jingzhou Central Hospital (Other); Wuhan University (Other); Wuhan Central Hospital (Other); Central Command General Hospital (Unknown); Second Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other); Heze Municipal Hospital (Other); Qingdao Central Hospital (Other); Taian City Central Hospital (Other); Yantai Yuhuangding Hospital (Other); Zibo First Hospital (Other); Huashan Hospital (Other); Fudan University (Other); Ruijin Hospital (Other); Dongfang Hospital Affiliated to Tongji University (Other); Changhai Hospital (Other); Henan Provincial People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Taikang Xianlin Drum Tower Hospital (Unknown); Xinqiao Hospital of Chongqing (Other); The First People Hospital of Nantong City (Unknown); Wuxi People's Hospital (Other); The First People's Hospital of Changzhou (Other); The First People's Hospital of Yunnan (Other); People Hospital of Dali Bai Autonomous Prefecture (Unknown); First Affiliated Hospital of Kunming Medical University (Other); The Second Affiliated Hospital of Air Force Military Medical University (Unknown); The 306 Hospital of People's Liberation Army (Other); The Sixth Central Hospital of PLA (Unknown); Peking University Third Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); China Rehabilitation Research Center (Other Government); The Third People Hospital of Datong (Unknown); Dezhou People's Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: CJFH
Record Dates: First submitted 2021-03-28; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Nutritional Deficiency
Keywords: Nutritional Management; Respiratory Critically Ill Patients; Enteral Nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The important role of nutritional management in the treatment of ICU patients has been paid more and more attention. Reasonable nutritional management can improve the nutritional status of patients, reduce the risk of malnutrition, shorten the length of ICU stay, improve the quality of life of patients, and reduce the mortality of patients, thereby improving the prognosis. Many studies have investigated the nutritional status and implementation of ICU patients. It is generally believed that the nutritional status of ICU patients is not good, and the implementation of standardization needs to be improved.The data on the nutritional status and implementation of RICU patients in mainland China is rare. Therefore, the main purpose of this study is to investigate the implementation and compliance of nutritional support treatment for RICU patients in mainland China.

DETAILED DESCRIPTION:
Respiratory critically ill patients have their own disease metabolism and treatment methods. However, RICU medical staff generally do not pay enough attention to nutrition support treatment. The data on the nutritional status and implementation of RICU patients in China is rare. But the data plays an important role in carrying out nutrition-related research, formulating the goals of continuing education programs for nutrition support treatment, guiding the introduction of medical insurance policies and the revision of consensus. Therefore, the main purpose of this study is to investigate the implementation and compliance of nutritional support treatment for RICU patients in tertiary hospitals in mainland China, so as to lay the foundation for further relevant work.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >18 years
* the length of RICU stays >48 hours

Exclusion Criteria:

* patients aged ≤18 years
* the length of RICU stays ≤48 hours
* patients who were admitted to RICU due to or combined with severe trauma or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients admitted to RICU
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of enteral nutrition starting within 48 hours after ICU entry | 48 hours
  Proportion of enteral nutrition starting within 48 hours after ICU entry

SECONDARY OUTCOMES:
Nutritional status and risk of malnutrition on ICU admission | 48 hours
  To assess nutritional status and risk of malnutrition on ICU admission by NRS-2002 risk score and NUTRIC score
The proportion of subjects receiving>80% estimated energy target within 7 days after ICU entry | 7 days
  The proportion of subjects receiving>80% estimated energy target within 7 days after ICU entry
The proportion of enteral nutrition intolerance | 48 hours
  The proportion of enteral nutrition intolerance

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang X, Wang Y, Geng S, Liang Y, Gao F, Wang T, Zhang H, Fang J, Wang C, Gu X, Yang J, Cheng Z, Liu C, Lei W, Hu X, Luo H, Fan H, Zhang Y, Li G, Di Q, Xing L, Li Y, Tong J, Chen L, Sun W, Chen L, Wang S, Li S, Liu J, Qin H, Qiu X, Ma Z, Li Y, Zhao H, Liang R, Wang L, Gao P, Sang L, Li D, Hou P, Zhang X, Wang D, Zheng L, Hua F, Jiang J, Li X, Nie Q, Zhao H, Huang C, Ji Y, Yu H, Song L, Jin J, Li N, Qian W, Zeng J, Chen L, Sun J, He W, Guan S, Chai S, Hu S, Li G, Li J, Jiang H, Zhong X, Li J, Zhao J, Du W, Zhang J, Liu Z, van Zanten A, Tian Y, Cai Y, Zhan Q. Nutritional practices and impact of feeding adequacy on clinical outcomes in Chinese respiratory intensive care units patients: a prospective observational study (ORIENT study). Front Nutr. 2026 Jan 20;12:1719386. doi: 10.3389/fnut.2025.1719386. eCollection 2025. PMID 41640734